CLINICAL TRIAL: NCT02606370
Title: Effects of Unstable Shoes on Trunk Muscle Activity, Lumbar Spine Kinematics and Pain in Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Head of Medicine, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA
Record Dates: First submitted 2015-11-11; First posted 2015-11-17 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Low Back Pain
Keywords: Unstable Shoes;Trunk muscles;Lumbar lordosis;Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unstable shoes (Experimental): Wearing unstable shoes during 1 month
  Interventions: Other: Unstable shoe
- Control Group (No Intervention): Not Wearing unstable shoes

INTERVENTIONS:
Other: Unstable shoe — Wearing Unstable shoes during 1 month
  Arms: Unstable shoes

SUMMARY:
Aim: To compare trunk muscle activity, lumbar spine range of motion (ROM) and LBP during gait using an unstable shoe (Intervention group) and a conventional stable control shoe (Control Group).

Design: Randomized Controlled Trial. Setting: A Biomechanics laboratory. Population: Patients with Low Back Pain.

DETAILED DESCRIPTION:
Background: An unstable shoe was developed as a walking device to strengthen the lower extremity muscles and reduce joint loading. A large number of studies have reported increased electromyographic (EMG) activity throughout the gait cycle in most of the lower limb muscles, and significant kinematic changes in the lower extremity. However, no studies have investigated the effects of wearing (1 month) unstable shoes on 1) spine kinematics, 2) trunk muscle activity and 3) Low Back Pain (LBP) during gait in Patients with chronic LBP.

Aim: To compare trunk muscle activity, lumbar spine range of motion (ROM) and LBP during gait using an unstable shoe (Intervention group) and a conventional stable control shoe (Control Group).

Design: Randomized Controlled Trial. Setting: A Biomechanics laboratory. Population: Patients with Low Back Pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic LBP
* BMI < 30

Exclusion Criteria:

* Hernia
* Lower limb pathologies
* Previous experience with unstable shoes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Disability (assessed by Roland Morris Questionaire) | At 1 month

SECONDARY OUTCOMES:
EMG activity of trunk muscles | At baseline and at 1 month follow-up
Lumbar spine range of movement (sagittal plane) | At baseline and at 1 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: JF Lisón, Dr., Study Director — Cardenal Herrera University; Pablo Salvador-Coloma, Principal Investigator — Cardenal Herrera University
Locations (1):
- University CEU Cardenal Herrera, Moncada, Valencia, Spain

REFERENCES:
- [Result] Lison JF, Perez-Soriano P, Llana-Belloch S, Sanchez-Zuriaga D, Salvador-Coloma P. Effects of unstable shoes on trunk muscle activity and lumbar spine kinematics. Eur J Phys Rehabil Med. 2016 Aug;52(4):440-6. Epub 2015 Apr 9. PMID 25854301